CLINICAL TRIAL: NCT04807556
Title: The Alusti Test: Turkish Validity and Reliability Study of the "Functional Evaluation Scale of Physical Performance in the Geriatric Population".
Brief Title: The Alusti Test:Functional Evaluation Scale of Physical Performance in the Geriatric Population
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Other Study IDs: 004
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-09

CONDITIONS: Functional Assessment Scale of Physical Performance (Alusti Test) for the Geriatric Population

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Alusti Test — Physical and psychological functional conditions are key factors in the elderly population

SUMMARY:
With the Alusti Test, which is created by Josu Alustiza Navarro considering the existing tests, the physical performances of geriatricians with different levels and cognitive capacity are evaluated in a very short time and without tiring the patient. There are 2 versions, short and full. The short version is applicable to 100% of the large population, including "and cases of cognitive impairment. With the full version, it has nearly 85-90% applicability."

However, there is no study regarding the English version and validity reliability of the 'Alusti Test.

For this purpose, it is to investigate the English validity and reliability of the functional assessment scale of physical performance (Alusti Test) for the geriatric population and to provide a measurement tool to be used in the English literature to the sciences who want to work in this field.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 65,
* volunteering
* to be able to read and write
* To be able to read and write in Turkish

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Over the age of 65 geriatrics
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Alusti test | 5 minute
  Physical and psychological functional conditions are key factors in the elderly population. Many evaluation tools are available, but they cannot be applied to the whole geriatric population. The use Alusti Test is presented.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB). | 5 minute
  Short Physical Performance Battery (SPPB) is an assessment test used to examine gait, balance, strength, and endurance in elderly epidemiological studies and outpatient clinics. Its performance is divided into three subtests: a hierarchical balance assessment, a short usual gait speed test, and 5 Time Sit to Stand (5TSTS) test
TimedUp and Go (TUG). | 3 minutes
  It is a clinical assessment test widely used to assess balance and walking ability in elderly populations [19-21]. To perform this test, participants are observed and timed in seconds, while they rise from an armed chair of approximately 46cm seat height and 65 cm arm height, walk at their usual pace a distance of 3 meters towards a line marked on the floor, turn 180 degrees, walk back to the chair, and sit down
Mini-Mental State Examination (MMSE) | 3 minutes
  Cognitive status was assessed using the Mini-Mental State Examination (MMSE); MMSE scores were categorized into three levels (0-17, 18-23, and 24-30, indicating severe, mild, and no impairment, respectively).
Tinetti Test | 5 minutes
  The Tinetti test has been recommended and widely used in the elderly to assess mobility, balance and gait, and predict falls. D
Rivermead Mobility Index | 10 minute
  The Rivermead Mobility Index (RMI) is a hierarchical mobility scale used in neurological rehabilitation. It includes 15 items related to bed mobility, transfers, walking, stair use, and running. The RMI is presented in a questionnaire format with the examiner required to make one observation (standing unsupported >10 s). All items are rated in a yes/no format with positive responses scoring a 1 for a maximal RMI score of 15.
Barthel Index | 5 minute
  The Barthel index (BI) is a widely used observer-based instrument to measure physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Atıcı, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided